CLINICAL TRIAL: NCT01751438
Title: A Prospective, Multi-Institutional, Randomized, Phase II Trial of Best Systemic Therapy or Best Systemic Therapy (BST) Plus Definitive Treatment (Radiation or Surgery) of the Primary Tumor in Metastatic (M1) Prostate Cancer (PC)
Brief Title: Best Systemic Therapy or Best Systemic Therapy (BST) Plus Definitive Treatment (Radiation or Surgery)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0705; NCI-2013-00415 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate carcinoma; Metastatic; M1; Best Systemic Therapy; BST; Androgen deprivation therapy; Bilateral orchiectomy; Radiation; Radiation Therapy; External beam radiation therapy; External-beam radiotherapy; Xray therapy; XRT; Surgery
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Surgical Procedures, Operative; Radiotherapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best Systemic Therapy (BST) (Experimental): Group 1 will continue to receive best systemic therapy (BST). Questionnaire completion at 60 days, 12 weeks, and at end of treatment visit. It should take about 15 minutes to complete. Every 6 months after end-of-treatment visit, patient contacted by phone or e-mail and asked questions about how they are feeling. Each phone call should last about 5 minutes.
  Interventions: Other: Best Systemic Therapy (BST); Behavioral: Questionnaires; Other: Phone Call/Email
- Best Systemic Therapy (BST) + Surgery or Radiation Therapy (Experimental): Group 2 will receive best systemic therapy (BST) in addition to surgery to remove prostate or radiation therapy to the prostate. Treating physician will decide if surgery or radiation therapy is the best choice. Questionnaire completion at 60 days, 12 weeks, and at end of treatment visit. It should take about 15 minutes to complete. Every 6 months after end-of-treatment visit, patient contacted by phone or e-mail and asked questions about how they are feeling. Each phone call should last about 5 minutes.
  Interventions: Other: Best Systemic Therapy (BST) + Surgery or Radiation Therapy; Behavioral: Questionnaires; Other: Phone Call/Email

INTERVENTIONS:
Other: Best Systemic Therapy (BST) — Group 1 will continue to receive best systemic therapy (BST).
  Arms: Best Systemic Therapy (BST)
Other: Best Systemic Therapy (BST) + Surgery or Radiation Therapy — Group 2 will receive best systemic therapy in addition to surgery to remove prostate or radiation therapy to the prostate. Treating physician will decide if surgery or radiation therapy is the best choice.
  Arms: Best Systemic Therapy (BST) + Surgery or Radiation Therapy
Behavioral: Questionnaires — Questionnaire completion at 60 days, 12 weeks, and at end of treatment visit. It should take about 15 minutes to complete.
  Other Names: Surveys
Other: Phone Call/Email — Every 6 months after end-of-treatment visit, patient contacted by phone or e-mail and asked questions about how they are feeling. Each phone call should last about 5 minutes.

SUMMARY:
The goal of this clinical research study is to learn if treatment with standard systemic therapy (androgen deprivation therapy or bilateral orchiectomy) in combination with surgery or radiation therapy is more effective at controlling prostate cancer than standard systemic therapy alone. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups at 6 months (+/- 14 days) from starting standard systemic therapy. You will have an equal chance of being assigned to each group.

* If you are in Group 1, you will continue to receive standard of care systemic treatment.
* If you are in Group 2, you will receive standard of care systemic treatment in addition to surgery to remove your prostate or radiation therapy to the prostate. You and your treating physician will decide if surgery or radiation therapy is the best choice for you. Your treating physician will explain the surgery or radiation therapy and their risks to you in more detail, and you will be asked to sign a separate consent form for the procedure.

If the disease gets worse within the first 6 months of receiving standard systemic therapy, you will not be assigned to a study group. You may be able to continue receiving standard systemic therapy if your doctor thinks it is in your best interest. You may choose to participate in this study by allowing the study team to collect information about you at the following study visits described below: within 60 days of screening, end-of-treatment, and long-term followup.

Study Visits:

Within 60 days after screening:

* You will have a physical exam, including a digital rectal exam (DRE).
* You will be asked how well you are able to perform the normal activities of daily living (performance status).
* Blood (about 2-3 teaspoons) will be drawn for routine tests, to check your prostate-specific antigen (PSA) levels, and testosterone levels.
* Urine will be collected for routine tests.
* You will complete a questionnaire about how you are feeling. It should take about 15 minutes to complete.
* You will have a bone scan, 2 CT scans of your abdomen and pelvis, and a chest X-ray or a computed tomography (CT) scan of chest to check the status of the disease.
* You will have a endorectal Magnetic Resonance Imaging (MRI) scan of the prostate to check the status of the disease.

Every 12 weeks (+/- 14 days) while on study (starting at month 9):

* You will have a physical exam, including a DRE and any updates to your medical history will be recorded.
* You will be asked about any side effects you may have had.
* You will be asked about any drugs or treatments you may be receiving, including over-the-counter drugs, herbal remedies, vitamins, and/or supplements.
* Blood (about 2-3 teaspoons) will be drawn for routine tests, to check your liver function, and to measure PSA and testosterone levels.
* You will complete a questionnaire about how you are feeling. It should take about 15 minutes to complete.
* If the study doctor thinks it is needed, you will have CT/MRI imaging scans to check the status of the disease.

If you are not having side effects after the 12-month visit, you will be given a PSA kit so you can send in a sample to test your PSA level. You will need to have your blood (about 1 teaspoon) drawn at your local doctor's office or lab and mail the kit in, every 3 months. The package will be provided, but you will need to pay postage. You would still need to visit the clinic every 6 months. The study staff will tell you more about this.

Length of Treatment:

You may continue your participation in this study for as long as the doctor thinks it is in your best interest. You will be taken off the study treatment if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your active participation on the study will be over after the long-term follow-up phone calls/emails (described below).

End-of-Treatment Visit:

Within 14 days after your study treatment is stopped, the following tests and procedures will be performed:

* You will have a physical exam, including a DRE.
* You will be asked about any side effects you may have had.
* You will be asked about any drugs or treatments you may be receiving, including over-the-counter drugs, herbal remedies, vitamins, and/or supplements.
* Blood (about 2-3 teaspoons) will be drawn for routine tests, to check your liver function, and to measure PSA and testosterone levels.
* Urine will be collected for biomarker testing.
* You will complete a questionnaire about how you are feeling. It should take about 15 minutes to complete.
* If the study doctor thinks it is needed, you will have CT/MRI imaging scans to check the status of the disease.

Long-Term Follow-Up:

Every 6 months after your end-of-treatment visit for up to 10 years, you will be contacted by phone or e-mail, and you will be asked questions about how you are feeling. Each phone call should last about 5 minutes. If you are not able to be contacted by phone or email, the study doctor will review and record any updates to your medical record.

This is an investigational study. Using standard of care systemic treatment with surgery, and/or radiation therapy are both FDA approved and commercially available.

Up to 180 patients will take part in this multi-center study. Up to 180 patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients
2. 18 yrs and older
3. Histologically or cytologically proven prostate carcinoma
4. Documented evidence of M1 disease by AJCC (American Joint Committee on Cancer) staging by Bone scan, CT and/or MRI.
5. Androgen dependent disease measured by declining PSA and do not display signs of progression demonstrated by a rising PSA.
6. Treatment initiation with BST no longer than 6 months prior to randomization
7. ECOG PS 0 or 1
8. Life-expectancy based on comorbid conditions >2 years
9. Ability to understand and willingness to sign informed consent
10. Must be a candidate for surgery and/or radiation therapy

Exclusion Criteria:

1. Psychiatric or medical conditions which, in the opinion of the treating physician, would not allow the patient to undergo the proposed treatments safely.
2. Known brain metastasis
3. Small cell carcinoma of the prostate
4. Any laboratory abnormalities, which in the opinion of the investigator, may put the subject at risk if participating in the study. For example: AST + ACT > 2 upper limits of normal value; WBC < 2.0; Hgb < 7.0.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 60 days
  Primary endpoint is progression-free survival, defined as the time interval from the start of initial best systemic therapy (BST) treatment to the date of disease progression or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Brian F. Chapin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - UCSF University of California, San Francisco, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Vancouver Prostate Center, Vancouver, British Columbia, Canada

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org